CLINICAL TRIAL: NCT02037945
Title: 18F-Fluorocholine (18F-FCho) to Distinguish Necrosis From Recurrence in Brain Metastases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 13-199
Record Dates: First submitted 2014-01-14; First posted 2014-01-16 (Estimated); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Brain Metastases
Keywords: 18F-Fluorocholine (18F-FCho); Pet Scan; MRI; 13-199
MeSH Terms: conditions — Brain Neoplasms

ARMS (1):
- pts with brain mets going for surgery (Experimental): This study will enroll patients with brain metastases that are evolving after SRS who are scheduled to undergo surgical resection. Eligible patients will undergo an 18F-FCH PET study 1-to-7 days pre-operatively. Although no toxicity has been previously reported following 18F-FCH administration, patients will be contacted 1-3 days after their scan and asked whether they experienced any adverse effects. The patients who have a positive 18F-FCH PET study (in which there is visible focal "hot spots" (a focus of lesion/normal white matter ratio >1.4) of 18F-FCH) will undergo further evaluation and be administered a second administration oflower activity 18F-FCH at the time of surgery. The purpose of the second 18F-FCH administration in the operating room is to further elucidate the tissue distribution of 18F-FCH radioactivity with respect to the histopathology of the surgically resected tissue.
  Interventions: Procedure: 18F-FCH PET Scan

INTERVENTIONS:
Procedure: 18F-FCH PET Scan

SUMMARY:
The main purpose of this study is to determine the distribution of 18F Fluorocholine (18F-FCH) in the brain which can help distinguishing radiation-induced scarring from tumor regrowth. In addition, the study will measure levels of 18F-FCH in the blood and (if applicable) in the brain lesion tissue that is removed as part of the planned brain surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient and/or guardian is able to provide written informed consent prior to study registration
* Age ≥ 21 years old
* Evolving brain lesions post SRS requiring neurosurgical resection (whether for symptomatic control or to establish pathology)

Exclusion Criteria:

* Inability to undergo a MRI or PET scan (e.g., claustrophobia or metal implant)
* Pregnant or nursing female
* Unable to cooperate for PET/CT

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2022-12-08 (Actual); Study Completion 2022-12-08 (Actual)

PRIMARY OUTCOMES:
to distinguish radiation necrosis from progressive tumor | 1 year
  by comparing the PET imaging results to the surgical pathology

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Beal, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

DOCUMENTS (1):
  • Informed Consent Form (2014-10-14): https://cdn.clinicaltrials.gov/large-docs/45/NCT02037945/ICF_000.pdf